CLINICAL TRIAL: NCT04862351
Title: Effectiveness of Technology-assisted Interventions in Hybrid Cardiac Rehabilitation (TechCR) Among Coronary Heart Disease Patients
Brief Title: Effectiveness of TechCR Among CHD Patients
Acronym: TechCR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Mei Sin CHONG, Principal Investigator, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2020.621
Record Dates: First submitted 2021-04-07; First posted 2021-04-28 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Coronary Heart Disease
Keywords: technology-assisted interventions; hybrid cardiac rehabilitation; coronary heart disease
MeSH Terms: conditions — Coronary Disease | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: The eligible participants will be randomly assigned into either intervention group (IG) or control group (CG) in 1:1 ratio using the computerised permuted blocks, alternating block sizes of 4 or 6. Once the eligible participants have consented to participate and the baseline data is collected, they will be given an opaque sealed envelope prepared by an independent statistician (not involved in the research) with assignment information and group allocation specified in the envelope. According to Polit and Beck (2017), the risk of selection bias can be reduced through allocation concealment by shielding the researcher from knowing the next group allocation of an individual.
Who Masked: Outcomes Assessor
Masking Description: A single blinding will be implemented for the outcome assessor as the participants will not be able to be blinded due to the nature of the interventions. The participants will not be informed directly whether they are in the intervention group or control group but the information regarding the intervention will be stated in the Participant Information Sheet. Thus, the participants may know their group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TecHCR (Experimental): 12 weeks Hybrid between supervised exercise training and video call sessions Educational videos Dietary and exercise log
  Interventions: Behavioral: exercise training for TechCR; Behavioral: audio/video conference; Behavioral: educational video; Behavioral: Daily log
- Centre-based (Other): 12 weeks usual care provided by the centre-based, outpatient cardiac rehabilitation clinic Dietary and exercise log
  Interventions: Behavioral: Daily log; Behavioral: exercise training for centre-based

INTERVENTIONS:
Behavioral: exercise training for TechCR — 3 times of supervised exercise training at the centre-based, outpatient cardiac rehabilitation clinic
  Arms: TecHCR
Behavioral: audio/video conference — weekly audio/video conference
  Arms: TecHCR
Behavioral: educational video — weekly for 6 weeks, duration of video about 10-15 minutes
  Arms: TecHCR
Behavioral: Daily log — daily dietary and exercise log
Behavioral: exercise training for centre-based — 6 times of supervised exercise training
  Arms: Centre-based

SUMMARY:
During this ongoing pandemic, there is a crucial need for innovative approaches to deliver CR programmes other than frequent face-to-face sessions at the centre-based CR to reduce the number of times people come close in contact with others or gathering in large groups. This is a single setting, 2-arm parallel randomised clinical trial which aims to examine the effects of technology-assisted interventions in hybrid cardiac rehabilitation (TecHCR) among the coronary heart disease patients. Eligible participants will be randomly assigned into either intervention group (IG) or control group (CG) in 1:1 ratio using the computerised permuted blocks, alternating block sizes of 4 or 6. All participants will be followed up for three months and six months with data collection at baseline, (T0), three-month (T1) and six-month (T2) time points.

DETAILED DESCRIPTION:
In recent years, CR delivery platforms and approaches have been changing as technology has become an integral part of our daily lives. Some of the barriers to CR may be able to be tackled with the advancement of technology, as it provides an alternative to the traditional centre-based CR through virtual consultations and remote monitoring that may eliminate the hassle of face-to-face consultations, work and time conflicts. During this ongoing pandemic, there is a crucial need for innovative approaches to deliver CR programmes other than frequent face-to-face sessions at the centre-based CR to reduce the number of times people come close in contact with others or gathering in large groups.

The overall aim of this proposed study is to examine the effects of technology-assisted interventions in hybrid cardiac rehabilitation (TecHCR) among the coronary heart disease patients. The objectives are as followings:

1. to determine the effects of TecHCR on self-efficacy related to exercise;
2. to determine the effects of TecHCR on health promoting behaviours;
3. to determine the effects of TecHCR in adherence;
4. to determine the effects of TecHCR in exercise capacity;
5. to determine the effects of TecHCR on fasting low density lipoprotein (LDL), high density lipoprotein (HDL), total cholesterol, systolic blood pressure, diastolic blood pressure, body mass index and waist circumference;
6. to determine the effects of TecHCR anxiety and depression.

With the attrition rate of 20%, a total of 160 eligible participants with 80 per group will be recruited. The control group receives usual care including outpatient medical follow-up with the cardiologists and dietician counselling before hospital discharge. Then, the participants will have their first follow-up by the physicians in cardiac rehabilitation clinic and followed by monthly follow-up. Subsequently, they will have weekly, centre-based supervised exercise training by physiotherapist and follow-up with occupational therapist for 12 weeks. In addition of the usual care of outpatient medical follow-ups and dietary education, the intervention group will receive 3 times supervised exercise in the centre, weekly upload of CR education (audio-visual video) on WhatsApp for six weeks (Week 1 to Week 6). The prescribed exercise will then be continued at home with a pedometer as the "cue to action" to be worn by the participant; he or she will be required to upload the data daily to the web app on the smartphone. Participants will also receive a weekly audio/video-conferencing follow-up (Week 1 to Week 12). The outcome measures include Socio-demographic and Clinical Data, Bandura's exercise self efficacy scale (ESE), Health Promoting Lifestyle Profile II (HPLP II), adherence referring to the attendance to 12 weeks (supervised exercise training) for CG, and attendance (3 times supervised exercise training) and upload of exercise data (for 9 weeks) to web app for IG; and 12-week assessment for both groups, exercise capacity by Exercise Stress Test measuring the metabolic equivalents METs) and Hospital Anxiety and Depression Scale (HADS). The data entry and analysis will be performed using the IBM Social Package Statistical Software (SPSS) version 26.0 with a p value < 0.05 will be consider significant of the result.

ELIGIBILITY:
Inclusion Criteria:

1. adults ≥ 18 years old;
2. patients with documented acute myocardial infarction, treated with thrombolysis, angioplasty or revascularisation surgery;
3. patients who own a mobile phone with internet access;
4. patients who have at least completion of primary school education;
5. understand English or Malay language;
6. patients who will return home for living after hospital discharge;
7. patients who are medically stable and referred to CR programme and able to give informed consent to participate in this study.

Exclusion Criteria:

1. patients who are participating in other studies;
2. patients who will undergo any repeat cardiac or other procedure in next 12 months;
3. patients with comorbidities such as dementia, impaired hearing or vision or psychiatric illness which may affect the ability to participate in the CR programme;
4. patients with pre-existing mobility problems which prevent them from exercising

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2021-02-26 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2023-10-31 (Actual)

PRIMARY OUTCOMES:
self-efficacy related to exercise (Bandura's Exercise Self-efficacy) | Baseline (T0) - at 0 week, before initiation of interventions
  Using Bandura's Exercise Self-efficacy to determine the effects of TecHCR on self-efficacy related to exercise before intervention (baseline)
self-efficacy related to exercise (Bandura's Exercise Self-efficacy) | post intervention (T1) - at 12 weeks after initiation of interventions
  Using Bandura's Exercise Self-efficacy to determine the effects of TecHCR on self-efficacy related to exercise post intervention (at 3-month)
self-efficacy related to exercise (Bandura's Exercise Self-efficacy) | 6-month post intervention (T2) - at 36 weeks after initiation of interventions
  Using Bandura's Exercise Self-efficacy to determine the effects of TecHCR on self-efficacy related to exercise 3-month post intervention (T2) (at 6 month)

SECONDARY OUTCOMES:
behavioural outcomes (Health-promoting Lifestyle Profile II) | Baseline (T0) - at 0 week, before initiation of interventions
  Using Health-promoting lifestyle Profile II to determine the effects of TecHCR on health promoting behaviours
behavioural outcomes (Health-promoting Lifestyle Profile II) | post intervention (T1) - at 12 weeks after initiation of interventions
  Using Health-promoting lifestyle Profile II to determine the effects of TecHCR on health promoting behaviours
behavioural outcomes (Health-promoting Lifestyle Profile II) | 6-month post intervention (T2) - at 36 weeks after initiation of interventions
  Using Health-promoting lifestyle Profile II to determine the effects of TecHCR on health promoting behaviours
psychological outcomes (Hospital Anxiety and Depression Scale) | Baseline (T0) - at 0 week, before initiation of interventions
  Using Hospital Anxiety and Depression Scale to determine the effects of TecHCR on anxiety and depression
psychological outcomes (Hospital Anxiety and Depression Scale) | post intervention (T1) - at 12 weeks after initiation of interventions
  Using Hospital Anxiety and Depression Scale to determine the effects of TecHCR on anxiety and depression
psychological outcomes (Hospital Anxiety and Depression Scale) | 6-month post intervention (T2) - at 36 weeks after initiation of interventions
  Using Hospital Anxiety and Depression Scale to determine the effects of TecHCR on anxiety and depression
fasting low density lipoprotein (LDL), high density lipoprotein (HDL), total cholesterol (from laboratory blood test result) | Baseline (T0) - at 0 week, before initiation of interventions
  to determine the effects of TecHCR on fasting low density lipoprotein (LDL), high density lipoprotein (HDL), total cholesterol (mmol/L)
fasting low density lipoprotein (LDL), high density lipoprotein (HDL), total cholesterol (from laboratory blood test result) | post intervention (T1) - at 12 weeks after initiation of interventions
  to determine the effects of TecHCR on fasting low density lipoprotein (LDL), high density lipoprotein (HDL), total cholesterol (mmol/L)
fasting low density lipoprotein (LDL), high density lipoprotein (HDL), total cholesterol (from laboratory blood test result) | 6-month post intervention (T2) - at 36 weeks after initiation of interventions
  to determine the effects of TecHCR on fasting low density lipoprotein (LDL), high density lipoprotein (HDL), total cholesterol (mmol/L)
systolic and diastolic blood pressure (using blood pressure monitoring device) | Baseline (T0) - at 0 week, before initiation of interventions
  to determine the effects of TecHCR on systolic and diastolic blood pressure
systolic and diastolic blood pressure (using blood pressure monitoring device) | post intervention (T1) - at 12 weeks after initiation of interventions
  to determine the effects of TecHCR on systolic and diastolic blood pressure
systolic and diastolic blood pressure (using blood pressure monitoring device) | 6-month post intervention (T2) - at 36 weeks after initiation of interventions
  to determine the effects of TecHCR on systolic and diastolic blood pressure
Body Mass Index (BMI) (weight in kilogrammes*height in metres^2) | Baseline (T0) - at 0 week, before initiation of interventions
  to determine the effects of TecHCR on BMI
Body Mass Index (BMI) (weight in kilogrammes*height in metres^2) | post intervention (T1) - at 12 weeks after initiation of interventions
  to determine the effects of TecHCR on BMI
Body Mass Index (BMI) (weight in kilogrammes*height in metres^2) | 6-month post intervention (T2) - at 36 weeks after initiation of interventions
  to determine the effects of TecHCR on BMI
Waist circumference (measured by measuring tape in centimetres) | Baseline (T0) - at 0 week, before initiation of interventions
  to determine the effects of TecHCR on waist circumference
Waist circumference (measured by measuring tape in centimetres) | post intervention (T1) - at 12 weeks after initiation of interventions
  to determine the effects of TecHCR on waist circumference
Waist circumference (measured by measuring tape in centimetres) | 6-month post intervention (T2) - at 36 weeks after initiation of interventions
  to determine the effects of TecHCR on waist circumference

CONTACTS AND LOCATIONS:
Overall Officials: Mei Sin Chong, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- University Malaya Medical Centre, Kuala Lumpur, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chong MS, Sit JWH, Choi KC, Suhaimi A, Jiang Y, Chair SY. The Effects of a Technology-Assisted Hybrid Cardiac Rehabilitation (TecHCR) Program for Adults With Coronary Heart Disease: A Randomized Controlled Trial. Worldviews Evid Based Nurs. 2025 Dec;22(6):e70092. doi: 10.1111/wvn.70092. PMID 41457512
- [Derived] Chong MS, Sit JWH, Choi KC, Suhaimi A, Chair SY. A Theory-Based, Technology-Assisted Intervention in a Hybrid Cardiac Rehabilitation Program for Patients with Coronary Heart Disease: A Feasibility Study. Asian Nurs Res (Korean Soc Nurs Sci). 2023 Aug;17(3):180-190. doi: 10.1016/j.anr.2023.06.004. Epub 2023 Jun 22. PMID 37355035